CLINICAL TRIAL: NCT05012475
Title: Assessing the Effectiveness of Customized Computer Activities on Reducing Stereotypies and Improving Independent Upper Extremity Motor Skills in Persons with Rett Syndrome
Brief Title: Measuring Impact of Computer Gaming on Arm Use in Rett Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: International Rett Syndrome Foundation Rettsyndrome.org (Unknown)
Responsible Party: Principal Investigator, Pamela Diener, Professor, Georgetown University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0656
Record Dates: First submitted 2021-08-04; First posted 2021-08-19 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Rett Syndrome
Keywords: enrichment; sensory stimulation; motor recovery; upper extremity function
MeSH Terms: conditions — Rett Syndrome

STUDY DESIGN:
Intervention Model Description: Investigators accept individuals with Rett syndrome who meet the inclusion criteria that requires functional arm range of motion, understanding of cause and effect and a diagnosis of Rett syndrome.
Masking Description: No masks needed as no direct contact will take place. This study is designed to be entirely virtual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participants (Experimental): The study involves a pre-intervention phase (4 weeks long), followed by a cause and effect training phase (1 week long), followed by an intervention phase (12 weeks long), and ending with a post-intervention phase (4-weeks long) for a total of 5-6 months from start to finish.
  Interventions: Behavioral: Modified Virtual Reality Gaming

INTERVENTIONS:
Behavioral: Modified Virtual Reality Gaming — Investigators customize each gaming session based on the motivators and interests of each participant. The intervention facilitates independent hand separations (minimizing stereotypies) and encourages independent arm/hand movement that serves to activate or control the computer-generated activities.

SUMMARY:
Using a tele-research approach, we will recruit, enroll, guide and support carers and participants to engage in computer based activities (modified virtual reality) with the primary outcome of reducing stereotypies and increasing independent arm and hand use and secondary outcome of improving quality of living. Because of our virtual approach, we are able to recruit from multiple countries and all states and territories of the USA.

DETAILED DESCRIPTION:
Early in life, individuals with Rett syndrome lose purposeful use of their hands and engage in handwringing and handmouthing stereotypies. It is important to pursue interventions that may facilitate the development and sustained use of arms/hands for productive involvement in daily needs that ultimately improve quality of life. Investigators plan to use a tele-research approach to assist caregivers and the participants in playing customized computer generated games that require independent and sustained hand separations and initiated and sustained movement patterns to control the modified virtual reality activity that serves as our intervention. Customization of the games and activities used will require collaboration with the caregivers of each participant to ensure that the level of motivation and interest of the participant matches the game/activities used. Brightly colored wristbands will be worn on each participant's wrist during the one-hour long intervention in which they will be involved 3 days per week for ~12 weeks. These wrist bands will be detected by the software we developed. As the participants move their arms, our software will detect these position changes and activate the computer-based activities. At 5 different points in the study investigators will test for changes in independent reaching abilities that may result from exposure to the intervention. Specifically, investigators will assess the impact of the intervention on minimizing hand stereotypies and improving the amount and quality of independent arm function. At the start and end of the study, investigators will also assess the impact the intervention had on activities of daily living, and therefore quality of life, via three goals developed in collaboration with the family/caregiver of the participant. Due to the virtual nature (tele-research) of the study, investigators aim to recruit 10-12 participants from multiple countries. Once enrolled, each participant will remain involved for up to 5-6 months. Since all activities are hand selected for each participant in collaboration with the caregivers, risks of involvement in this study are low. Investigators anticipate that this intervention will improve motor planning abilities for arm use and reduce stereotypies.

ELIGIBILITY:
Inclusion Criteria:

* Rett syndrome,
* Understanding of cause and effect,
* Functional range of motion of arms to complete the movements needed to control the games.

Exclusion Criteria:

* no competing orthopedic or neuromuscular diagnosis that impacts shoulder movements

Ages: 4 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
functional Reach Test | To measure change, this test is administered (repeated) 5 times during the 5 month study: Day 1 (baseline); Day 32 (start of wk long training); Day 40 (after one wk training session); Day Day 130 (end of 12 wk intervention); Day 160 (post-intervention).
  Investigators will video record all testing sessions so that the video can be viewed slow motion or frame by frame to count hand separations, number of reaches, time of sustained reaches, and sustained hand separations.

SECONDARY OUTCOMES:
Goal Attainment Scale (GAS) | To measure change, this test is administered on Day 1 (Baseline) and repeated at Day 120 (end of intervention phase)
  In collaboration with the parents/carers, investigators will create three goals specific for each participant that relate to study aims and improving quality of daily living.
Functional Range of Motion (FROM) | To assess if a change in FROM occurs during the study, this test is administered on Day 1 (Baseline) and repeated at Day 120 (Post-intervention)
  Assess range of shoulder and hand motion at start and at end of study to be sure that shoulder mobility is unchanged and/or not impacting the required motions for the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Georgetown University School of Medicine, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] McAmis NE, Foreman MH, Himmelrich MD, Diener PS and Engsberg JR. Development of a Method to Use a Color Tracker for Motor Therapy for Individuals with Rett Syndrome. SM J Pediatr. 2017; 2(2): 1012.
- [Background] Mraz KM, Amadio G, Diener P, Eisenberg G, Engsberg JR. Improving upper extremity motor skills in girls with rett syndrome using virtual reality. J of Intellect Disabil - Diagnosis and Treatment, 2016, 4(3):142-151.
- [Background] Mraz, K, Eisenberg G, Diener P, Amadio G, Foreman MH, Engsberg JR. The Effects of Virtual Reality on the Upper Extremity Skills of Girls with Rett Syndrome: A Single Case Study. J of Intellect Disabil- Diagnosis and Treatment. 2016, 4(3):152-9.